CLINICAL TRIAL: NCT03066310
Title: Detection of Bladder Cancer Using Urinary Cell-free DNA and Cellular DNA
Brief Title: Urine-DNA Biomarkers in Detecting Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Hunan Cancer Hospital (Other); Hunan Provincial People's Hospital (Other); Second People's Hospital of Hunan (Other)
Responsible Party: Sponsor
Other Study IDs: XYURO002
Record Dates: First submitted 2017-02-20; First posted 2017-02-28 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer; Biomarker; Diagnosis; Urine
Keywords: Bladder cancer; Urine; DNA biomarker; Diagnosis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Voided urine samples were collected prior to the cystoscopy and stored at 4 ℃，within 12 hours after collection ,urine samples were processed in paticipant laboratories. Blood samples was collected. Tissue samples was collected( optional).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnosed Urinary Bladder Cancers: Patients who are being monitored for bladder cancer will be the experimental group to test the urine-DNA by next generation sequencing for bladder cancer biomarkers
  Interventions: Diagnostic Test: Next generation sequencing
- Non-Urinary Bladder Cancers: Patients being treated for gross hematuria will provide a negative control to provide data from testing by next generation sequencing for biomarkers in patients being treated for other diseases.
  Interventions: Diagnostic Test: Next generation sequencing

INTERVENTIONS:
Diagnostic Test: Next generation sequencing — The obtained DNA from the urine, blood and tumor (optional) will be tested by next generation sequencing for each arm.

SUMMARY:
DNA biomarkers in urine are important diagnostic and prognostic indicators for bladder cancer. Many genetic alterations have been identified in the urinary DNA. However, not all bladder tumors harbor mutations in the most commonly altered oncogenes. Thus, to reach satisfactory sensitivity and specificity a new diagnostic test should include multiple biomarkers. The investigators will conduct a prospective evaluation of a panel of mutations in urine-DNA test for the detection of urothelial bladder carcinoma in patients with gross hematuria for cystoscope.

DETAILED DESCRIPTION:
Urinary DNA representative of the tumour genome provide a promising resource as a liquid biopsy for non-invasive genomic profiling of urothelial bladder cancers. Voided urine samples will be collected prior to cystoscopy. Cell free DNA and cellular DNA will both be extracted and analyzed. A blood sample will be taken. In patients with bladder wall findings suspicious of cancer, a bladder wall biopsy will be taken and submitted for histopathology examination, according to clinical standard practice. Next generation sequencing will be applied and hotspots mutations in DNA from urine, blood and tumor. Logistic regression was used to analyze the association between predictor variables and bladder cancer. The investigators will confirm a couple of common mutations occured in urine-DNA and blood-derived DNA simultaneously and verify the specificity and sensitivity of individual variance or mutation combinations to establish an predictive model with optimal robustness in diagnosis of bladder cancer. Moreover, external consistency test will be performed on subsequent patients collection.

ELIGIBILITY:
Inclusion Criteria:

* patients with gross hematuria or other clinical sympton suspected of bladder cancer.
* male or female patients aged >= 18 years.
* available tumor tissue, urine and blood sample.
* signed informed consent form.

Exclusion Criteria:

* prior diagnosis of cancer except bladder cancer
* age under 18 years
* individuals unwilling to sign the IRB-approved consent form
* comorbidities that would prohibit or make serial urine collection and cystoscopy examine difficult or impossible.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients diagnosed with suspected bladder cancer in Xiangya Hospital of Central South University from February of 2017 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
sensitivity of urinalysis by Urine-DNA test | through study completion, an average of 8 months
  number of patients "declared positive" with the Urine-DNA test among the patients actually suffering from bladder carcinoma
specificity of urinalysis by Urine-DNA test | through study completion, an average of 8 months
  number of patients "declared negative" with the Urine-DNA test among the patients without bladder carcinoma
Identification of positive urine-DNA test results with the next generation sequencing | through study completion, an average of 8 months
  Identification of presence of positive urine-DNA test results with the designed panel.
Identification of urine-DNA mutations with the next generation sequencing to create an diagnosis algorithm. | through study completion, an average of 8 months
  Identification of presence or absence of the mutations in urine-DNA with the next generation sequencing to create an idiagnosis algorithm

SECONDARY OUTCOMES:
sensitivity of blood DNA test | through study completion, an average of 8 months
  number of patients "declared positive" with the blood-DNA test among the patients actually suffering from bladder carcinoma
specificity of blood DNA test | through study completion, an average of 8 months
  number of patients "declared negative" with the blood DNA test among the patients without bladder carcinoma
comparison of the sensitivity of the urine DNA versus blood DNA test | through study completion, an average of 8 months
  number of patients "declared positive" with the urine DNA test versus patients "declared positive" with the blood DNA test.
comparison of the specificity of the urine DNA versus blood DNA test | through study completion, an average of 8 months
  number of patients "declared negative" with the urine DNA test versus patients "declared negative" with the blood DNA test.

CONTACTS AND LOCATIONS:
Overall Officials: Long Wang, M.D., Ph.D, Study Chair — Xiangya Hospital of Central South Univeristy
Locations (1):
- Xiangya Hospital of Central South Univeristy, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided